CLINICAL TRIAL: NCT00084240
Title: A Phase 2/3, Randomized, Comparative, Double Blind Trial Of Azithromycin Plus Chloroquine Versus Sulfadoxine-Pyrimethamine Plus Chloroquine For The Treatment Of Uncomplicated, Symptomatic Falciparum Malaria In Southeast Asia
Brief Title: Azithromycin Plus Chloroquine Versus Sulfadoxine-Pyrimethamine Plus Chloroquine For The Treatment Of Uncomplicated, Symptomatic Falciparum Malaria In Southeast Asia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661123
Record Dates: First submitted 2004-06-09; First posted 2004-06-11 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Azithromycin/Chloroquine
Drug: Sulfadoxine-Pyrimethamine/Chloroquine

SUMMARY:
The primary objective is to confirm the hypothesis that azithromycin (optimal dose once daily for three days) plus chloroquine is non-inferior to sulfadoxine-pyrimethamine plus chloroquine for the treatment of uncomplicated, symptomatic malaria due to P. falciparum.

DETAILED DESCRIPTION:
The trial was terminated prematurely 2 June 2005 due to the inability to recruit the planned number of subjects. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Females and males >=18 years of age with uncomplicated, symptomatic malaria as indicated by the presence of both of the following: a.) Blood smears positive for Plasmodium falciparum asexual parasitemia between 1000 -100,000 parasites/mL b.) Fever or history of fever (>= 38.5 C/101.2 F rectal or tympanic; >= 37.5 C/99.5 F axillary or >= 38 C/100.4 F oral) within the prior 24 hours
* Serum glucose >= 60 mg/dL (by fingerstick or peripheral blood collection)
* Positive rapid diagnostic test (Binax NOW ICT) for P. falciparum
* Women of childbearing potential must have a negative urine gonadotropin prior to entry into the study and must agree to use adequate contraception during the entire study

Exclusion Criteria:

* Severe or complicated malaria including subjects with any of the following: a.) Impaired consciousness, seizures or abnormal neurologic exam b.) Jaundice c.) Respiratory distress d.) Persistent vomiting e.) Hematuria, as reported by the patient f.) Parasite density > 100,000 parasites/mL g.) Presence of non-falciparum species on microscopy
* Pregnant or breast-feeding women
* History of allergy to or hypersensitivity to azithromycin or any macrolide, sulfonamides, pyrimethamine, or chloroquine
* Known history of blood dyscrasias (e.g., megaloblastic anemia, agranulocytosis, aplastic anemia, thrombocytopenia, leukopenia, neutropenia, hemolytic anemia)
* History of epilepsy or psoriasis
* History of treatment with any antimalarial drug (chloroquine, quinine, mefloquine, Malarone, SP, artemisinin compounds) or antibacterial with known antimalarial activity (macrolides, doxycycline, clindamycin) within 2 weeks prior to enrollment into the study
* Known or suspected cardiovascular, hepatic or renal abnormality that in the opinion of the Investigator would place the subject at increased risk to participate in the study. The following findings are specific exclusions: a.) serum creatinine > 2.0 x ULN b.) ALT and/or AST > 3 x ULN
* Inability to swallow oral medication in tablet form
* Treatment with other investigational drugs within 30 Days prior to enrollment into the study
* Alcohol and/or any other drug abuse
* Requirement to use medication during the study that might interfere with the evaluation of the study drug (nelfinavir, digoxin, ergot alkaloids, terfenadine, cyclosporine, hexobarbital and phenytoin)
* Specific systemic diseases or other medical conditions that would interfere with the evaluation of the therapeutic response or safety of the study drug
* Inability to comprehend and/or unwillingness follow the study protocol
* Intentions to leave the vicinity of the trial site in the next 42 days
* Prior participation in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-03; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
parasite clearance

SECONDARY OUTCOMES:
tolerability and safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer